CLINICAL TRIAL: NCT00149396
Title: A Phase I/II, Open-label Study to Evaluate the Safety and Anti-tumor Effects of NV1020 Administered Repeatedly Via Hepatic Artery Infusion Prior to Second-line Chemotherapy, in Patients With Colorectal Adenocarcinoma Metastatic to the Liver
Brief Title: Safety & Efficacy of NV1020 in Colorectal Cancer Metastatic to the Liver
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MediGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT1030
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Cancer; Liver Neoplasms
Keywords: Colorectal cancer metastases to liver; Colorectal Cancer; Colorectal Carcinoma; Colorectal Tumors; Colorectal Neoplasms; Rectum Cancer; Rectum tumors; Rectum carcinoma; Colon cancer; Colon tumors; Colon carcinoma; Rectum Neoplasms; Colon Neoplasms; Liver Neoplasms; Hepatic Neoplasms; Liver Tumors; Liver cancer; Hepatic Cancer; Hepatic tumors; metastatic to the liver
MeSH Terms: conditions — Colorectal Neoplasms; Liver Neoplasms; Rectal Neoplasms; Colonic Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Safety and antitumor effects of NV1020 (Experimental): Stage 1: Four escalating dose cohorts of NV1020 3x10^6 pfu, 1x10^7 pfu, 3x10^7 pfu, and 1x10^8 pfu administered via hepatic artery infusion, over 10 minutes and repeated every 1-2 weeks for 4-8 weeks followed by 2 cycles of chemotherapy.
  Stage 2: Expansion of one dose cohort from Stage 1 of optimal NV1020 dose administered via hepatic artery infusion, over 10 minutes and repeated every 1-2 weeks for 4-8 weeks followed by 2 cycles of chemotherapy.
  Interventions: Drug: NV1020

INTERVENTIONS:
Drug: NV1020 — NV1020 dose levels: 3x10^6, 1x10^7, 3x10^7, and 1x10^8 plaque forming units, administered via hepatic artery infusion, over 10 minutes and repeated every 1-2 weeks for 4-8 weeks

SUMMARY:
This study is an open-label study. It has two stages. Stage 1 is a dose escalation phase of the study to determine and evaluate the safety and tolerability of repeated treatments with a genetically engineered herpes simplex virus NV1020 administered locoregionally to the liver.

Stage 2 is to evaluate the dose found in Stage 1 to be "optimally tolerated". Stage 2 is to assess the efficacy of the optimally tolerated dose of NV1020 by itself and in combination with second-line chemotherapy.

Assignment to Stage 1 or Stage 2 of the study is determined by when the patient enters the study.

DETAILED DESCRIPTION:
This study is designed to evaluate the effects of repeated treatments with NV1020, prior to second-line chemotherapy, and to determine an appropriate dose level of NV1020 in a multiple dose regimen for later Phase II studies.

Sequential, open-label cohort dose escalation of NV1020 (stage 1) followed by an expansion of one selected dose cohort (stage 2).

Study results will be reviewed periodically by an independent DSMB who will approve each cohort dose escalation.

During the dose escalation stage, 3 cohorts of patients (3 in each) will be treated with 4 fixed doses of NV1020, with the dose level increasing for successive cohorts. A patient will be observed for a minimum of 7 days after the first NV1020 infusion before the next patient in the same cohort is given NV1020. The first patient in the next higher dose cohort will receive NV1020 no earlier than 14 days after the last patient in the prior cohort has finished NV1020 infusions. One additional cohort (half log higher increment) may be approved by the DSMB, if considered necessary to define MTD. Dose-limiting toxicity will be determined using NCI CTC criteria and a suitable dose level for later evaluation will be selected.

In the second stage of the study, the dose cohort considered to show the best therapeutic index will be expanded by the addition of 18 further patients. For all patients in this study, investigational treatment with NV1020 will be followed by a minimum of two cycles of second-line therapy using anti-neoplastic drugs approved by the FDA for colorectal cancer and selected by the investigator.

All patients will be followed up periodically until death. Permission for autopsy will be sought.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign a written informed consent (includes willingness to avoid physical intimacy during and for 2 weeks post NV1020 treatment)
2. 18 years or more of age
3. Colorectal adenocarcinoma histologically confirmed within one year prior to enrollment in the study
4. Liver dominant metastases (CT-measurable lesions with less than 50% total liver involvement), histologically confirmed
5. Failed conventional chemotherapy for metastatic disease (e.g. tumors no longer responding to 5-FU/leucovorin in combination with irinotecan or oxaliplatin with or without one monoclonal antibody)
6. Candidate for additional chemotherapy (and/or experimental anti-cancer therapy, if this is the only remaining treatment option)
7. Karnofsky Performance Status 70% or greater
8. Life expectancy greater than or equal to 4 months, based on the investigator's opinion
9. Seropositive for herpes simplex virus-1 (HSV-1)
10. Fecund females: negative for pregnancy test (urine or serum)
11. Effective double-barrier contraception for a minimum of 2 months following final infusion of NV1020

Exclusion Criteria:

1. Dominant extrahepatic disease, including cerebral metastases, significant malignant ascites or other extrahepatic metastases that are symptomatic, in critical locations or otherwise likely to confound NV1020 evaluations, in the opinion of the investigator
2. Seronegative for HSV-1
3. Significant active/unstable non-malignant disease or laboratory test (hematology and chemistry) results that meet any of the following:

   * White blood cell count (WBC) less than or equal to 3 x 10e3/mm3
   * Absolute neutrophil count (ANC) less than or equal to 1.5 x 10e3/mm3
   * Platelets less than or equal to 100,000/mm3
   * Hemoglobin (Hgb) less than or equal to 9.0 g/dL
   * Prothrombin time/partial thromboplastin time (PT/PTT) > upper limit of normal (ULN)
   * Serum creatinine > 2.0 mg/dL
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 times ULN or total bilirubin > 1.5 times ULN
   * Alkaline phosphatase > 2.5 times ULN
4. Chemotherapy < 4 weeks prior to the first NV1020 infusion (mitomycin or nitrosurea < 6 weeks)
5. Immunotherapy < 6 weeks prior to the first NV1020 infusion
6. Radiotherapy (external or internal) to the liver
7. Major surgery (excluding pump placement and cholecystectomy) ≤ 2 weeks prior to the first NV1020 infusion but the subject must be clinically stable. Pump placement and cholecystectomy ≤ 1 week prior to the first NV1020 infusion but the subject must be clinically stable
8. Female who is pregnant or nursing
9. Patients wishing to conceive within 2 months after the last infusion of NV1020
10. Any investigational agent administered less than or equal to 4 weeks prior to NV1020 infusion
11. Acute HSV infection requiring systemic antiviral therapy or history of serious HSV infection (e.g., ocular, encephalitic, etc.)
12. Active viral hepatitis (evidence for infection with hepatitis A, B or C viruses)
13. Known infection with HIV
14. Known hypersensitivity to any component of the NV1020 formulation
15. History of, or current, bleeding or coagulation disorder
16. History of significant hepatic fibrosis, cirrhosis, or hemachromatosis
17. History of malignancy other than colorectal cancer, within 5 years prior to start of study participation, with the exception of in situ cervical or skin carcinoma
18. Active severe infection and any other concurrent disease or medical conditions that are likely to interfere with the study, as judged by the investigator
19. Systemic corticosteroid administration < 4 weeks prior to starting NV1020 treatment
20. Prior treatment with NV1020 or other putative oncolytic viruses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-07; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hoda Tawfik, PhD, Study Director — MediGene
Locations (5):
- United States (5):
  - University of California, San Diego, San Diego, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Pittsburgh Cancer Center, Pittsburgh, Pennsylvania
  - University of Vanderbilt, Nashville, Tennessee
  - Mary Crowley Medical Research Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sze DY, Iagaru AH, Gambhir SS, De Haan HA, Reid TR. Response to intra-arterial oncolytic virotherapy with the herpes virus NV1020 evaluated by [18F]fluorodeoxyglucose positron emission tomography and computed tomography. Hum Gene Ther. 2012 Jan;23(1):91-7. doi: 10.1089/hum.2011.141. Epub 2011 Oct 14. PMID 21895536

RESULTS

PARTICIPANT FLOW:
Groups:
- NV1020: Escalating doses of NV1020: 3x10^6, 1x10^7, 3x10^7, 1x10^8
Period: Overall Study
Arm/Group | NV1020
Started | 32
Completed NV1020 Therapy | 29
Completed NV1020 and Chemotherapy | 9
Completed | 9
Not Completed | 23
Not completed — Death | 15
Not completed — Withdrawal by Subject | 1
Not completed — Subject noncompliance | 2
Not completed — other treatment | 5

BASELINE CHARACTERISTICS:
Arm/Group | NV1020
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 21
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 29
  African American | 1
  Asian | 1
  Hispanic | 1
Carcinoembryonic Antigen (CEA) Level at Screening [Mean (Standard Deviation); unit: ng/mL] | 175.5 (517.4)
Prior Chemotherapy [Number; unit: participants] | 32
Karnofsky Performance Status (KPS) [Number; unit: participants] — The KPS was rated as follows:
  100 - Normal, no complaints, no evidence of disease; 90 - Able to carry on normal activity; minor signs or symptoms of disease; 80 - Normal activity with effort; some signs or symptoms of disease
  participants
    KPS 100 | 14
    KPS 90 | 17
    KPS 80 | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events and Dose Limiting Adverse Events
Description: Incidence of adverse events for all patients (N=32); Overall incidence ≥20%; Adverse events listed by Medical Dictionary for Regulatory Activities (MedDRA) Preferred Term
Time Frame: From start of treatment through 12 months after completion of treatment
Measure: Number; unit: percentage of participants
Groups:
- All Patients: All patients in study
Arm/Group | All Patients
Number analyzed (Participants) | 32
percentage of participants
  Dose limiting adverse events | 0
  Nausea | 69
  Abdominal pain | 47
  Diarrhea | 44
  Vomiting | 41
  Abdominal pain upper | 25
  Constipation | 22
  Pyrexia | 94
  Chills | 56
  Fatigue | 56
  Edema peripheral | 22
  Back pain | 34
  Headache | 41
  Anemia | 41
  Neutropenia | 22
  Rash | 28
  Hypokalemia | 22
  Insomnia | 22

2. Secondary Outcome: Mean Change From Baseline in Serum Carcinoembryonic Antigen (CEA) After Administration of NV1020 and 2 Cycles of Chemotherapy
Time Frame: Screening (baseline), Chemo visit 1, Chemo visit 2, Follow-up Visit 1 (1 week after end of treatment), Follow-up Visit 2 (+6M), Follow-up Visit 3 (+9M), Follow-up Visit 4 (+12M)
Population: Number of participants analyzed decreases through the follow-up visits. Thus the "Number of Participants Analyzed" indicated here refer to the number at baseline.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Dose Cohort 1: NV1020 Dose 3x10^6 pfu (Stage 1)
- Dose Cohort 2: NV1020 Dose 1x10^7 pfu (Stage 1)
- Dose Cohort 3: NV1020 Dose 3x10^7 pfu (Stage 1)
- Dose Cohort 4: NV1020 Dose 1x10^8 pfu (Stages 1 and 2)
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4
Number analyzed (Participants) | 3 | 3 | 4 | 22
ng/mL
  Mean Baseline CEA | 1814.4 (3105.2) | 161.0 (235.1) | 121.6 (230.3) | 181.7 (373.3)
  Mean Change - Chemo visit 1 | 869.6 (1489.9) | 96.0 (106.1) | 8.6 (17.0) | 165.6 (410.5)
  Mean Change - Chemo visit 2 | 17.9 (13.2) | 194.4 (212.8) | -0.6 (NA) — N=1 for this timepoint | 98.2 (254.1)
  Mean Change - Follow-up 1 | -353.9 (628.8) | 615.6 (867.5) | 5.4 (5.8) | 97.0 (334.1)
  Mean Change - Follow-up 2 | 6995.9 (12110.6) | 134.7 (NA) — N=1 for this timepoint | 1.8 (3.5) | 97.3 (311.9)
  Mean Change - Follow-up 3 | NA (NA) — N=0 for this timepoint | NA (NA) — N=0 for this timepoint | 16.5 (NA) — N=1 for this timepoint | -52.3 (94.9)
  Mean Change - Follow-up 4 | NA (NA) — N=0 for this timepoint | NA (NA) — N=0 for this timepoint | -1.7 (NA) — N=1 for this timepoint | 290.9 (447.8)

3. Secondary Outcome: Liver Tumor Response After Administration of NV1020 Followed by Chemotherapy, Determined by Radiological (Computed Tomography [CT] Scan) Assessment
Description: Maximum percentage changes in tumor diameter after administration of NV1020 followed by chemotherapy as measured by CT scan and Modified Response Evaluation Criteria in Solid Tumors (RECIST) assessment
Time Frame: Screening (baseline), Chemo visit 1, Follow-up visits 1 (1 week post end of treatment), 2 (+6M), 3 (+9M), 4 (+12M)
Measure: Number; unit: percentage
Groups:
- Stage 1: Escalating doses of NV1020: 3x10^6 pfu, 1x10^7 pfu, 3x10^7 pfu, 1x10^8 pfu
- Stage 2: Optimal dose from Stage 1: 1x10^8 pfu
Arm/Group | Stage 1 | Stage 2
Number analyzed (Participants) | 13 | 19
percentage
  Patient 101 | 22.70 | NA — This patient not in Stage 2 of study
  Patient 102 | 41.76 | NA — This patient not in Stage 2 of study
  Patient 103 | 18.85 | NA — This patient not in Stage 2 of study
  Patient 201 | 36.91 | NA — This patient not in Stage 2 of study
  Patient 202 | 21.55 | NA — This patient not in Stage 2 of study
  Patient 203 | 25.00 | NA — This patient not in Stage 2 of study
  Patient 301 | 4.92 | NA — This patient not in Stage 2 of study
  Patient 302 | 24.55 | NA — This patient not in Stage 2 of study
  Patient 303 | 10.74 | NA — This patient not in Stage 2 of study
  Patient 304 | 2.68 | NA — This patient not in Stage 2 of study
  Patient 401 | -24.51 | NA — This patient not in Stage 2 of study
  Patient 402 | -5.36 | NA — This patient not in Stage 2 of study
  Patient 403 | -7.98 | NA — This patient not in Stage 2 of study
  Patient 801 | NA — This patient not in Stage 1 of study | 5.45
  Patient 802 | NA — This patient not in Stage 1 of study | 35.89
  Patient 803 | NA — This patient not in Stage 1 of study | -35.56
  Patient 804 | NA — This patient not in Stage 1 of study | 21.43
  Patient 805 | NA — This patient not in Stage 1 of study | 11.41
  Patient 806 | NA — This patient not in Stage 1 of study | 18.90
  Patient 807 | NA — This patient not in Stage 1 of study | 29.98
  Patient 808 | NA — This patient not in Stage 1 of study | 16.77
  Patient 809 | NA — This patient not in Stage 1 of study | 30.00
  Patient 810 | NA — This patient not in Stage 1 of study | 57.67
  Patient 811 | NA — This patient not in Stage 1 of study | -1.93
  Patient 812 | NA — This patient not in Stage 1 of study | -19.05
  Patient 813 | NA — This patient not in Stage 1 of study | 25.29
  Patient 814 | NA — This patient not in Stage 1 of study | 114.29
  Patient 815 | NA — This patient not in Stage 1 of study | 9.38
  Patient 816 | NA — This patient not in Stage 1 of study | 12.20
  Patient 817 | NA — This patient not in Stage 1 of study | 3.30
  Patient 818 | NA — This patient not in Stage 1 of study | -11.19
  Patient 819 | NA — This patient not in Stage 1 of study | -24.18

4. Secondary Outcome: Pharmacodynamic Effects of NV1020: NV1020 Neutralizing Antibody Titer Assay
Description: Mean change from baseline in NV1020 neutralizing antibody titer by dose cohort
Time Frame: Screening, Chemo Visit 1, Follow-up Visits 1 (1 week post end of treatment), 2 (+6M), 3 (+9M), 4 (+12M)
Measure: Mean (Standard Deviation); unit: antibody titer
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4
Number analyzed (Participants) | 3 | 3 | 4 | 22
antibody titer
  Mean Baseline Neutralizing Antibody | 282.7 (96.4) | 1242.7 (1585.2) | 1006.6 (844.6) | 334.2 (309.1)
  Mean Change - Chemotherapy Visit 1 | 1341 (914) | 1061 (1430) | 4926 (1444) | 3481 (2251)
  Mean Change - Follow-up Visit 1 | 1231 (1382) | 950 (1344) | 2154 (473) | 2389 (1736)
  Mean Change - Follow-up Visit 2 | 824 (622) | 1152 (NA) — N=1 for this timepoint | 1887 (1133) | 1292 (1245)
  Mean Change - Follow-up Visit 3 | NA (NA) — N=0 for this timepoint | NA (NA) — N=0 for this timepoint | 450 (NA) — N=1 for this timepoint | 1029 (863)
  Mean Change - Follow-up Visit 4 | NA (NA) — N=0 for this timepoint | NA (NA) — N=0 for this timepoint | -543.1 (NA) — N=1 for this timepoint | 403 (374)

5. Secondary Outcome: Time to Disease Progression; Survival Time
Description: Progression assessed from CT and PET measurements and is determined as an increase of greater than or equal to 25% in the sum of the products of perpendicular diameters of all tumors, or the appearance of any new lesion.
Time Frame: Progression: Chemo visit 1, FU1 (1 week post treatment), FU2 (+6M), FU3 (+9M), FU4 (+12M); Survival: death of patient
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 1 | Stage 2
Number analyzed (Participants) | 13 | 19
months
  Median time to progression | 3.5 [2.8 to 6.9] | 6.4 [2 to 8.9]
  Median survival time | 12.4 [9.6 to 15.0] | 11.6 [8.3 to 20.7]

6. Primary Outcome: NV1020 Pharmacokinetics - Presence of NV1020 in Body Fluids/Skin
Description: Number of patients with NV1020 detected in saliva, skin, and/or mucosal surfaces; Analysis by polymerase chain reaction (PCR)
Time Frame: Daily for 2 weeks after the first and last NV1020 infusions
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 32
participants | 0

7. Primary Outcome: Clinical Laboratory Safety - Hematology
Description: Number of patients with clinically significant hematology laboratory abnormalities by NV1020 dose cohort (Post baseline)
Time Frame: Screening; after each NV1020 infusion; +7h, +24h, and +72h after NV1020 infusion; each chemotherapy visit; +3d, +7d, +14d after each chemo visit; 1 week after end of treatment
Measure: Number; unit: participants
Groups:
- Dose Cohort 2: NV1020 Dose: 1x10^7 pfu (Stage 1)
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4
Number analyzed (Participants) | 3 | 3 | 4 | 22
participants
  Absolute neutrophil count (x10^3/uL) | 1 | 0 | 0 | 0
  Basophils (%) | 0 | 0 | 0 | 1
  Eosinophils (%) | 0 | 0 | 0 | 2
  Hematocrit (%) | 0 | 1 | 0 | 3
  Hemoglobin (g/dL) | 0 | 1 | 0 | 3
  Lymphocytes (%) | 1 | 0 | 0 | 1
  Monocytes (%) | 1 | 1 | 0 | 1
  Neutrophils (bands) (%) | 1 | 0 | 0 | 0
  Neutrophils (segs) (%) | 1 | 0 | 0 | 2
  Platelets (x10^3/uL) | 0 | 0 | 0 | 3
  Red blood cells (x10^6/uL) | 0 | 0 | 0 | 1
  White blood cells (x10^3/uL) | 1 | 0 | 0 | 7

8. Primary Outcome: Clinical Laboratory Safety - Chemistry
Description: Number of patients with post-baseline clinically significant laboratory chemistry abnormalities by NV1020 dose cohort
Time Frame: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4
Number analyzed (Participants) | 3 | 3 | 4 | 22
participants
  Alkaline Phosphatase (U/L) | 2 | 2 | 0 | 8
  ALT (SGPT) (U/L) | 0 | 0 | 0 | 6
  AST (SGOT) (U/L) | 1 | 0 | 0 | 6
  Bicarbonate (mmol/L) | 0 | 0 | 0 | 1
  BUN (mg/dL) | 0 | 1 | 0 | 0
  Calcium (mg/dL) | 0 | 0 | 0 | 0
  Chloride (mmol/L) | 0 | 0 | 0 | 1
  Creatinine (mg/dL) | 1 | 1 | 0 | 0
  Glucose (mg/dL) | 1 | 1 | 0 | 0
  Potassium (mmol/L) | 0 | 1 | 0 | 4
  Sodium (mmol/L) | 0 | 0 | 0 | 0
  Total Bilirubin (mg/dL) | 1 | 0 | 0 | 5
  YGT/GGT (U/L) | 2 | 2 | 0 | 5

9. Primary Outcome: Clinical Laboratory Safety - Coagulation
Description: Number of patients with post-baseline clinically significant laboratory coagulation abnormalities by NV1020 dose cohort
Time Frame: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4
Number analyzed (Participants) | 3 | 3 | 4 | 22
participants
  C-reactive Protein (mg/dL) | 1 | 1 | 0 | 6
  D-dimer (ug/mL) | 2 | 1 | 0 | 6
  Fibrinogen (ug/mL) | 2 | 0 | 0 | 4
  INR | 0 | 0 | 0 | 0
  Prothrombin Time (PT) (sec) | 0 | 0 | 0 | 3
  Partial Thromboplastin Time (PTT) (sec) | 1 | 0 | 0 | 3

10. Secondary Outcome: Pharmacodynamic Effects of NV1020: Serum Cytokines (INF Gamma)
Description: Median change from baseline of Interferon (INF) gamma 8 hours post NV1020 infusion (Visits 1, 3, 5, 7)
Time Frame: Baseline, after each NV1020 infusion (Visit 1, Visit 3, Visit 5, Visit 7)
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4
Number analyzed (Participants) | 3 | 3 | 4 | 22
pg/mL
  Median Baseline INF gamma | 1.1 [0.6 to 1.9] | 0.9 [0.6 to 1.7] | 0.7 [0.6 to 1.3] | 0.6 [0.6 to 15.0]
  Median Change - Visit 1 (post 8 hr) | 5.8 [0.1 to 6.0] | 0.5 [-1.1 to 0.5] | 4.7 [3.0 to 6.0] | 22.9 [0.0 to 169.4]
  Median Change - Visit 3 (post 8 hr) | 7.7 [2.9 to 42.1] | 0.8 [-1.1 to 6.3] | 36.0 [15.9 to 111.4] | 51.8 [0.2 to 433.4]
  Median Change - Visit 5 (post 8 hr) | 2.5 [1.5 to 3.5] | 0.2 [-0.8 to 4.0] | 10.3 [9.7 to 64.4] | 18.8 [1.3 to 281.4]
  Median Change - Visit 7 (post 8 hr) | 1.3 [0.3 to 3.3] | -0.3 [-1.1 to 3.9] | 7.6 [4.3 to 13.0] | 18.1 [1.4 to 327.8]

11. Secondary Outcome: Pharmacodynamic Effects of NV1020: Serum Cytokines (IL-6)
Description: Median change from baseline of Interleukin-6 (IL-6) 8 hours post NV1020 infusion (Visits 1, 3, 5, 7)
Time Frame: Baseline, after each NV1020 infusion (Visit 1, Visit 3, Visit 5, Visit 7)
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4
Number analyzed (Participants) | 3 | 3 | 4 | 22
pg/mL
  Median Baseline IL-6 | 6.9 [4.2 to 8.3] | 11.0 [6.5 to 12.0] | 15.5 [3.7 to 31.0] | 6.2 [1.6 to 169.0]
  Median change - Visit 1 (post 8 hr) | 1.7 [-4.8 to 27.8] | 6.0 [0.0 to 19.0] | 16.5 [3.8 to 57.0] | 32.1 [-0.4 to 497.2]
  Median change - Visit 3 (post 8 hr) | 29.8 [16.1 to 194.7] | 3.0 [2.0 to 13.5] | 50.2 [34.0 to 475.0] | 60.6 [1.7 to 989.0]
  Median change - Visit 5 (post 8 hr) | 12.1 [8.8 to 26.7] | 14.5 [8.0 to 49.0] | 63.0 [17.3 to 102.0] | 32.2 [2.4 to 371.0]
  Median change - Visit 7 (post 8 hr) | 34.7 [19.1 to 44.8] | 8.5 [8.0 to 49.0] | 11.3 [10.0 to 62.0] | 43.0 [8.0 to 433.0]

12. Secondary Outcome: Pharmacodynamic Effects of NV1020: Serum Cytokines (TNF-alpha)
Description: Median change from baseline of tumor necrosis factor (TNF-alpha) 8 hours post NV1020 infusion (Visits 1, 3, 5, 7)
Time Frame: Baseline, after each NV1020 infusion (Visit 1, Visit 3, Visit 5, Visit 7)
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Dose Cohort 3 | Dose Cohort 4
Number analyzed (Participants) | 3 | 3 | 4 | 22
pg/mL
  Median Baseline TNF-alpha | 1.8 [0.6 to 2.9] | 2.0 [1.6 to 2.2] | 2.5 [1.8 to 4.9] | 1.3 [0.6 to 3.6]
  Median change - Visit 1 (post 8 hr) | 0.2 [-8.0 to 3.8] | 1.4 [0.2 to 4.1] | -0.2 [-2.5 to 0.6] | 2.4 [-0.9 to 6.6]
  Median change - Visit 3 (post 8 hr) | 3.6 [0.2 to 7.1] | 0.4 [0.0 to 1.5] | 2.3 [1.3 to 3.9] | 5.9 [0.3 to 22.0]
  Median change - Visit 5 (post 8 hr) | 2.3 [1.0 to 3.3] | 1.3 [-0.7 to 1.4] | 1.8 [1.1 to 2.2] | 5.5 [0.9 to 14.0]
  Median change - Visit 7 (post 8 hr) | 2.2 [0.9 to 2.7] | 1.5 [-0.8 to 2.4] | 0.8 [0.7 to 5.4] | 5.7 [1.4 to 11.3]

ADVERSE EVENTS:
Time Frame: 3 years, 11 months (First subject enrolled to last subject completed)
Description: *Serious adverse events exclude those which were deemed to be unrelated to NV1020
Arm/Group | NV1020
Serious Adverse Events (participants affected / at risk) | 5/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NV1020 (N=32)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NV1020 (N=32)
Nausea (Gastrointestinal disorders) | 22 (50)
Abdominal pain (Gastrointestinal disorders) | 15 (27)
Diarrhoea (Gastrointestinal disorders) | 14 (29)
Vomiting (Gastrointestinal disorders) | 13 (30)
Abdominal pain upper (Gastrointestinal disorders) | 8 (10)
Constipation (Gastrointestinal disorders) | 7 (7)
Abdominal distension (Gastrointestinal disorders) | 6 (6)
Abdonimal tenderness (Gastrointestinal disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 4 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Flatulence (Gastrointestinal disorders) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Pyrexia (General disorders) | 30 (111)
Chills (General disorders) | 18 (41)
Fatigue (General disorders) | 18 (36)
Edema peripheral (General disorders) | 7 (9)
Asthenia (General disorders) | 3 (4)
Chest pain (General disorders) | 3 (3)
Pain (General disorders) | 3 (3)
Disease progression (General disorders) | 2 (2)
Edema (General disorders) | 2 (2)
Temperature intolerance (General disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (19)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (6)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 13 (20)
Dizziness (Nervous system disorders) | 4 (5)
Hypoaesthesia (Nervous system disorders) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 13 (24)
Neurtopenia (Blood and lymphatic system disorders) | 7 (9)
Leukopenia (Blood and lymphatic system disorders) | 2 (4)
Lymphopenia (Blood and lymphatic system disorders) | 2 (15)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 9 (10)
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 (3)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (3)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (3)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (14)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (6)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminaenemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2)
Herpes simplex (Infections and infestations) | 3 (3)
Bronchitis (Infections and infestations) | 2 (2)
Oral candidiasis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Insomnia (Psychiatric disorders) | 7 (9)
Depression (Psychiatric disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 3 (3)
Confusional state (Psychiatric disorders) | 2 (2)
Hypertension (Vascular disorders) | 5 (5)
Hypotension (Vascular disorders) | 5 (9)
Haematoma (Vascular disorders) | 4 (4)
Weight decreased (Investigations) | 5 (7)
Aspartate aminotransferase increased (Investigations) | 3 (6)
Gamma-glutamyltransferase increased (Investigations) | 3 (6)
Fibrin D dimer increased (Investigations) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (4)
Jaundice (Hepatobiliary disorders) | 2 (2)
Incision site complication (Injury, poisoning and procedural complications) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 2 (4)
Tachycardia (Cardiac disorders) | 4 (4)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No